CLINICAL TRIAL: NCT02003911
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Azithromycin in Children Hospitalized With Acute Asthma Exacerbations
Brief Title: Azithromycin for Children Hospitalized With Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-05-187
Record Dates: First submitted 2013-11-21; First posted 2013-12-06 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma; Acute asthma exacerbation; Pediatric; Azithromycin; Macrolide; Length of Stay; Hospital Medicine
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin suspension (Experimental): Azithromycin suspension at 10mg/kg/dose (max 500mg)
  Once daily for 3 days
  Interventions: Drug: Azithromycin
- Placebo suspension (Placebo Comparator): Same volume as active drug
  Once daily for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin suspension (200mg/5mL)
  Arms: Azithromycin suspension
Drug: Placebo
  Arms: Placebo suspension

SUMMARY:
Asthma is a chronic lung condition in children, and often requires hospitalization for acute exacerbations. Azithromycin has been used successfully in other chronic lung diseases, including cystic fibrosis. Despite limited clinical evidence, some pediatricians use azithromycin in children hospitalized with asthma, citing either treatment of atypical pathogens or its proposed anti-inflammatory properties. This study proposes a clinical trial to determine if azithromycin will shorten length of stay in children hospitalized with acute asthma exacerbations.

DETAILED DESCRIPTION:
Asthma is a chronic lung condition that accounts for over 130,000 pediatric hospitalizations nationally at a cost of almost 1.4 billion dollars. Atypical pathogens have been implicated both in initiating asthma and triggering acute asthma exacerbations. Azithromycin, a macrolide antibiotic, is known to have antibacterial activity against atypical pathogens and gram positive bacteria. More recently, macrolides have been increasingly used and effective against gram negative bacteria and inflammation in the lungs of patients with chronic respiratory illnesses. This effect may be secondary to the immunomodulatory effects macrolides possess, in addition to their anti-bacterial effects. In long-term therapy with macrolides, patients with asthma have shown improved bronchiolar hyperreactivity, spirometry, symptoms, and quality of life. However, studies of short-term treatment in the acute setting and in children are limited. Some practitioners use azithromycin in the treatment of acute asthma, despite limited data.

The investigators propose a double-blind, randomized, placebo-controlled trial of azithromycin in children aged 4-12 years with persistent asthma hospitalized with acute asthma exacerbations. Children will be enrolled within 12 hours of admission and will be randomized to receive three days of either azithromycin or placebo suspension (10mg/kg/dose, max of 500mg). The primary outcome measure will be length of stay (LOS). Secondary outcome measures will include: days of school/work missed, readmission rates, return to medical care rates, recurrence of symptoms, and steroid courses. In the future, patients may also be approached to enroll in the "Mechanism Subset Study" a separate pilot and feasibility study which will require two blood samples and two nasal aspirate samples and will test for atypical pathogens, interleukin-8 levels, and neutrophil/eosinophil counts. The average length of stay for patients in this age range with asthma in 2011 at our institution was 3.0 days. The investigators will enroll to achieve a power of 80%, with an alpha of 0.05, which will require 107 patients in each group to detect a 16 hour (0.67 day) difference in the primary outcome, LOS. This study hypothesizes that azithromycin treatment in children hospitalized with acute asthma will decrease LOS.

ELIGIBILITY:
Inclusion Criteria:

* 4-12 years of age
* Admission diagnosis of asthma at the Children's Hospital at Montefiore
* History of persistent asthma (as defined by National Heart, Lung, and Blood Institute)

Exclusion Criteria:

* Concurrent bacterial infection requiring antibiotics
* Antibiotics received within previous 2 weeks
* Contraindication to azithromycin (including allergy to macrolides)
* Chronic lung disease other than asthma (including bronchopulmonary dysplasia, cystic fibrosis, bronchiectasis) or home oxygen requirement
* Immunodeficiency (primary or acquired)
* Chronic systemic steroid use
* Invasive or non-invasive mechanical ventilation required acutely as result of current asthma admission
* Significant cardiac co-morbidity (including hemodynamically significant cardiac disease or arrhythmia)
* Liver disease (hepatitis)
* Pregnancy
* Seizure disorder, currently on anti-epileptic medication)
* Receiving albuterol every 4 hours (q4h) at the time of enrollment
* Previous enrollment in study

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey C Douglas, MD, Principal Investigator — Montefiore Medical Center; Katherine O'Connor, MD, Study Director — Montefiore Medical Center; Diana S. Lee, MD, Study Director — Montefiore Medical Center; Alyssa H Silver, MD, Study Director — Montefiore Medical Center
Locations (1):
- The Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin Suspension: Azithromycin suspension at 10mg/kg/dose (max 500mg)
  Once daily for 3 days
  Azithromycin: Azithromycin suspension (200mg/5mL)
- Placebo Suspension: Same volume as active drug
  Once daily for 3 days
  Placebo
Period: Overall Study
Arm/Group | Azithromycin Suspension | Placebo Suspension
Started | 80 | 79
Completed | 78 | 72
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin Suspension | Placebo Suspension | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7.5 [5.3 to 9.4] | 7.1 [5.2 to 9.4] | 7.3 [5.2 to 9.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 51 | 53 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 56 | 111
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 33 | 73
  White | 11 | 14 | 25
  More than one race | 29 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0
PASS Score on enrollment [Mean (Standard Deviation); unit: Score on a scale] — PASS=Pediatric Asthma Severity Score
  Range 0 (best) - 6 (worst)
  Score at each time point is calculated by adding 3 elements:
  Wheeze (0= None/Mild, 1=Moderate, 2=Severe) Prolonged expiration (0= None/Mild, 1=Moderate, 2=Severe) Work of breathing (0= None/Mild, 1=Moderate, 2=Severe)
  Score on a scale | 2.35 (1.25) | 2.71 (1.29) | 2.53 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Hospital length of stay
Time Frame: Admission time to discharge time (average LOS is 3 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
days | 1.69 [1.33 to 2.48] | 1.86 [1.33 to 2.63]

2. Secondary Outcome: Readmission Rate
Description: Number of hospital readmissions for asthma at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 1 | 1

3. Secondary Outcome: School Missed
Description: Days of school missed by patient at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 0 | 0

4. Secondary Outcome: Work Missed
Description: Days of work missed by parent/guardian at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 0 | 0

5. Secondary Outcome: Emergency Room Visits
Description: Number of emergency room visits for asthma symptoms since discharge at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 6 | 7

6. Secondary Outcome: Physician Office Visits
Description: Number of physician office visits for asthma symptoms since discharge at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 7 | 5

7. Secondary Outcome: Recurrence of Asthma Symptoms
Description: Number of recurrences of asthma symptoms since discharge at telephone follow-up phone calls at 1-week and 1-month interval after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 18 | 23

8. Secondary Outcome: Steroid Courses
Description: Number of courses of oral steroids since discharge at telephone follow-up phone call 1-month after discharge
Time Frame: One month after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin Suspension | Placebo Suspension
Number analyzed (Participants) | 80 | 79
Participants | 8 | 11

9. Other Pre Specified Outcome: Routine Clinical Results and Symptoms
Description: Respiratory viral panel or rapid viral testing results (if obtained as part of medical care), chest x-ray results/lab results (if obtained as part of medical care), vital signs, medications received during admission, medication side effects (diarrhea, abdominal pain, vomiting, flatulence), transfer to intensive care unit, time of wean of beta-agonists (q3h and q4h), and asthma severity (PASS score) at time of enrollment.
Time Frame: One week after discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Azithromycin Suspension | Placebo Suspension
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/80 | 1/79
Other Adverse Events (participants affected / at risk) | 2/80 | 7/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin Suspension (N=80) | Placebo Suspension (N=79)
Transfer to PICU (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin Suspension (N=80) | Placebo Suspension (N=79)
Study Exit (Social circumstances) | 2 (2) | 7 (7)

LIMITATIONS AND CAVEATS:
1. Early termination and power of findings
2. Urban population may not be generalizable
3. High asthma severity of participants
4. Systemic steroids given during hospitalization
5. Antimicrobial role of azithromycin (Mechanism not studied)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02003911/Prot_SAP_000.pdf